CLINICAL TRIAL: NCT05549882
Title: A Novel Index to Predict the Failure of High-Flow Nasal Cannula in Patients with Acute Hypoxemic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of intensive care unit, Principal investigator, Clinical Professor, Southeast University, China
Other Study IDs: 2020ZDSYLL303-P02
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: High-flow nasal cannula; VOX （Volume-OXygenation）
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HFNC success group
  Interventions: Other: no intervention
- HFNC failure group: HFNC failure was defined as the subsequent need for invasive MV.

INTERVENTIONS:
Other: no intervention — no intervention
  Groups: HFNC success group

SUMMARY:
High-flow nasal cannula (HFNC) is increasingly used in patients with acute hypoxemic respiratory failure (AHRF) and has been shown to improve outcome in specific patient categories, including community acquired pneumonia and after extubation. Since HFNC failure and delayed intubation is associated with adverse clinical outcome, predicting HFNC failure is of clinical importance.

In patients with pneumonia and hypoxemic failure treated with HFNC, the ROX index (SpO2/FiO2 over respiratory rate), has been validated to predict the risk for endotracheal intubation. Increased respiratory rate, an important component of ROX, is used as an estimate for high respiratory drive, although it is well known that respiratory rate is insensitive to early changes in respiratory drive. Indeed, it has been shown that ROX worked best only after 12 hours after HFNC initiation. Earlier and more sensitive predictors of HFNC failure would be of clinical importance. Initially, elevated respiratory drive increases tidal volume (VT), but not respiratory rate. In addition, high VT has been linked to patient self-inflicted lung injury (P-SILI) and such may increase intubation rate in patients with AHRF. Taken together, from a physiological perspective, elevated TV may be a better predictor for HFNC failure compared to respiratory rate. Hence, we report an approach to measure VT generated by patients supported with HFNC and establish a novel index named VOX (Volume-OXygenation) based on VT to predict HFNC failure in patients with AHRF.

DETAILED DESCRIPTION:
Study design This is a multi-center prospective observational study performed over a 12-month period (from August 2022 to August 2023). The research premise was granted approval by the local Ethics Committee (2020ZDSYLL303-P02).

VOX index The VOX index was defined as the ratio of SpO2/FiO2 over VT. Investigators briefly interrupted HFNC (3 minutes) to measure VT using a mechanical ventilator (SV800, Mindray) in noninvasive ventilation (NIV) mode, as an "NIV test". Inspiratory support was set at 5 cmH2O and 5 cmH2O positive end-expiratory pressure level for all patients, and initial oxygen concentration was set as in HFNC. NIV was delivered through a face mask (ZS-MZ-A, Zhongshan Medical) and a double-pipe system, while minimizing leaks. In consideration of variations in VT, we recorded mean VT and respiratory rate for 1 minute under stable conditions.

Study protocol HFNC therapy was started within 15 minutes after recruitment and initiated with a 30-40 LPM minimum flow. Investigators adjusted FiO2 as suitable, targeting SpO2 of 92% or more, and the rate of flow set on the basis of the physician's decision. HFNC discontinuation and invasive mechanical ventilation (IMV) initiation were based on the intubation criteria defined in investigators clinical protocol, finial decisions were made by the physicians in charge, who were blinded to the VT during NIV test. HFNC failure was defined as a need for IMV, on account of NIV is not employed as the second line of ventila,ory support in the event of HFNC failure, in the participating units. Patient demographics, comorbidities, and chest radiographs prior to HFNC initiation were documented upon inclusion into the research analysis. The acute physiologic assessment and chronic health evaluation II (APACHE II) score along with the sequential organ failure assessment score (SOFA) were documented based on the highest scores in the 24h previous HFNC initiation. The time of HFNC onset was defined as 0h. Vital signs; HFNC settings including FiO2, flow rate, and temperature; clinical respiratory variables including RR, VT, and SpO2; diaphragmatic ultrasonography including diaphragmatic displacement, diaphragm thickness (tdi), and Δtdi% (was calculated as [tdi end-inspiration-tdi end-expiration/tdi end-expiration] ×100) were recorded at 0, 2, 6, 12, 18, and each 24h pre day following initiation of HFNC treatment until day 7. Variables of pulmonary gas exchange variables with the arterial line were documented at 0, 6, 12 and each 24h pre day following initiation of HFNC treatment until day 7 after initiation of HFNC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 years and 80 years of age
* RR > 25 breaths per minute
* PaO2/FiO2 ≤ 300 mmHg while breathing oxygen at a flow rate ≥ 10 liters per minute and PaCO2 ≤ 45 mmHg

Exclusion Criteria:

* Patients could strongly benefit from NIV (ie, patients with underlying chronic lung disease, or exacerbation of asthma, with cardiogenic pulmonary oedema, severe neutropenia (<500/mm3), or neuromuscular diseases such as myasthenia gravis and Guillain-Barre syndrome)
* Patients with severe shock, defined as a vasopressor dose> 0.3 μg/kg per min norepinephrine-equivalent to maintain SBP > 90 mmHg
* Patients with impaired consciousness with a GCS ≤ 12
* Patients with an urgent need for intubation (ie, respiratory or cardiac arrest, severe hypoxemia defined as PaO2/FiO2 < 50mmHg despite maximum oxygen support)
* Patients with contraindication to NIV (ie, unresolved vomiting, upper airway obstruction, hematemesis, recent major esophageal and upper abdominal surgery, or severe facial trauma) and HFNC (ie, epistaxis, nasal obstruction or acceptance of nasal surgery), intubated for diagnostic or therapeutic procedures (fiberoptic bronchoscopy or surgery), and patients with a 'do not resuscitate or intubate' order

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU due to AHRF and treated with HFNC (Optiflow™, Fisher & Paykel, New Zealand) were screened for enrollment.
Sampling Method: Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
HFNC failure | within 7 days
  HFNC failure was defined as a need for IMV, on account of NIV is not employed as the second line of ventilatory support in the event of HFNC failure, in the participating units

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, School of Medicine Southeast University Nanjing, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No